CLINICAL TRIAL: NCT05996718
Title: Improving Care Through Improv: Promoting Mastery in the Moment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Candace Kemp, Professor, Georgia State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P30AG064200 (NIH); DBSR-11114 (Other: NIA CROMS); P30AG064200 (NIH)
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Caregiver Burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Informal Caregivers of Persons Living with Dementia (Experimental): Participants will receive the training program, "Improving Care through Improv." This involves four weekly 2-hour in-person training sessions.
  Interventions: Behavioral: Training program pilot

INTERVENTIONS:
Behavioral: Training program pilot — This intervention for informal caregivers consists of training that will introduce participants to improvisational (improv) theatre and teach its core communication skills.

SUMMARY:
The goals of this clinical trial are to: 1) refine the training program, "Improving Care though Improv;" and 2) test the program for its influence self-perceived caregiving mastery (i.e., how persons assess their ability to provide care) among informal caregivers of persons living with moderate dementia. Forty-three informal caregivers will be involved in testing the training program. These individuals will be assigned to groups of between 8 to12 caregivers and take part in weekly 2-hour sessions held over a 4-week period. These caregivers will be taught improvisational (improv) theater skills, which involves being in the moment, self-awareness, and responsiveness to others. This group also will be asked to answer surveys questions about themselves and the person receiving care at three timepoints and invited to provide feedback on their training experiences.

ELIGIBILITY:
Inclusion Criteria:

* Actively engaged in the care of community-dwelling persons living with moderate dementia (4 or 5 on a 7-point dementia-staging scale) who is not likely to be institutionalized within the next 6 months
* Able to attend at least 3 of the 4 in-person sessions
* Ability to communicate in English

Exclusion Criteria: Potential participants were excluded if they did not meet the above criteria or anticipated moving their person to a skilled nursing facility within the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candace L Kemp, PhD, Principal Investigator — Georgia State Univeristy
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be made available to qualified researchers through a data sharing agreement that is consistent with NIH data sharing policies, as well as policies and practices established by the Roybal Center for Dementia Caregiving Mastery at Emory University. The data to be collected include common data elements, including the Caregiver Mastery Scale developed by Pearlin and colleagues, as well as demographic characteristics. Although these data will be de-identified prior to release for sharing, there remains a possibility of deductive disclosure of participants with unusual characteristics. Therefore, this data sharing agreement will require: 1) a commitment only to use the data for research purposes and not to identify any individual participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroy or return the data after analyses are completed.
Time Frame: Study data will be made available no later than the on-line publication date of the main findings from the final dataset.
Access Criteria: Researchers must qualify and enter into a data sharing agreement. The agreement requires: 1) a commitment only to use the data for research purposes and not to identify any individual participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroy or return the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Groups:
- Caregivers: Caregiver of a person living with dementia participating in the Improving Care through Improv intervention. During the intervention, participants attended four 2-hour weekly in-person group classes designed to enhance caregiver mastery and improve well-being among family members and friends providing care to someone living with dementia.
Period: Overall Study
Arm/Group | Caregivers
Started | 43
Completed Month 1 Assessment | 42
Completed | 40
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Caregivers
Number analyzed (Participants) | 43
Age, Continuous [Mean (Full Range); unit: Years] | 58.87 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 31
  More than one race | 1
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants] — This study was conducted in Atlanta, Georgia, USA.
  Participants
    United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Pearlin Mastery, Loss, and Competence: Caregiver Competence Subscale
Description: 4-item Likert-type scale; scores range from 4 to 16 with higher scores indicating greater feelings of competence.
Time Frame: at baseline, upon training completion (Week 4), and three months post baseline.
Population: Forty-three caregivers began the study; 42 completed the survey at Month 1; 40 completed the month 3 survey.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 43
Score on a scale
  Baseline | 11.10 (2.31)
  Month 1: number analyzed (Participants) | 42
  Month 1 | 11.63 (2.07)
  Month 3: number analyzed (Participants) | 40
  Month 3 | 11.93 (2.06)

2. Secondary Outcome: Perceived Stress Scale
Description: 14-item Likert-type scale. Scores range from 0 to 56 with higher scores indicating greater stress.
Time Frame: at baseline, upon training completion (Week 4), and three months post baseline.
Population: Forty-three caregivers began the study; 42 completed the survey at Month 1; 40 completed the month 3 survey.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 43
Score on a scale
  Baseline | 26.25 (8.43)
  Month 1: number analyzed (Participants) | 42
  Month 1 | 26.65 (9.45)
  Month 3: number analyzed (Participants) | 40
  Month 3 | 23.10 (8.16)

3. Secondary Outcome: Center for Epidemiological Studies-Depression Scale
Description: 20-item Likert-type scale. Scores range from 0 to 60 with higher scores indicating greater depression.
Time Frame: at baseline, upon training completion (Week 4), and three months post baseline.
Population: Forty-three caregivers began the study; 42 completed the survey at Month 1; 40 completed the month 3 survey.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 43
Score on a scale
  Baseline | 14.83 (9.30)
  Month 1: number analyzed (Participants) | 42
  Month 1 | 14.78 (9.45)
  Month 3: number analyzed (Participants) | 40
  Month 3 | 12.98 (9.40)

4. Secondary Outcome: State-Trait Anxiety Inventory
Description: 20-item Likert-type scale. Scores range from 20 to 80 with higher scores indicating greater anxiety.
Time Frame: at baseline, upon training completion (Week 4), and three months post baseline.
Population: Forty-three caregivers began the study; 42 completed the survey at Month 1; 40 completed the month 3 survey.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 43
Score on a scale
  Baseline | 36.15 (10.27)
  Month 1: number analyzed (Participants) | 42
  Month 1 | 35.38 (11.09)
  Month 3: number analyzed (Participants) | 40
  Month 3 | 34.85 (11.62)

5. Secondary Outcome: Zarit Burden Inventory
Description: 22-item scale with 4-point Likert scale responses. Scores range from 0 to 88 with higher scores indicating greater burden.
Time Frame: at baseline, upon training completion (Week 4), and three months post baseline.
Population: Forty-three caregivers began the study; 42 completed the survey at Month 1; 40 completed the month 3 survey.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 43
Score on a scale
  Baseline | 61.95 (16.32)
  Month 1: number analyzed (Participants) | 42
  Month 1 | 61.63 (15.19)
  Month 3: number analyzed (Participants) | 40
  Month 3 | 59.68 (16.43)

6. Secondary Outcome: Revised Memory and Behavioral Problems Checklist - FREQUENCY
Description: 24-item scale with 4-point Likert scale responses. Scores range from 0 to 96 with higher scores indicating greater behavioral expressions observed by caregivers among persons living with dementia.
Time Frame: at baseline, upon training completion (Week 4), and three months post baseline.
Population: Forty-three caregivers began the study; 42 completed the survey at Month 1; 40 completed the month 3 survey.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 43
Score on a scale
  Baseline | 37.20 (14.21)
  Month 1: number analyzed (Participants) | 42
  Month 1 | 36.55 (11.99)
  Month 3: number analyzed (Participants) | 40
  Month 3 | 38.05 (13.78)

7. Secondary Outcome: Quality of Life-Alzheimer's Disease Scale
Description: 13 items with a 4-point Likert scale. Scores range from 13 to with 52 with higher scores indicating greater quality of life among persons living with dementia
Time Frame: at baseline, upon training completion (Week 4), and three months post baseline.
Population: Forty-three caregivers began the study; 42 completed the survey at Month 1; 40 completed the month 3 survey.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 43
Score on a scale
  Baseline | 27.85 (5.15)
  Month 1: number analyzed (Participants) | 42
  Month 1 | 27.88 (4.20)
  Month 3: number analyzed (Participants) | 40
  Month 3 | 27.63 (5.16)

8. Secondary Outcome: Revised Memory and Behavioral Problems Checklist - REACTION
Description: as for outcome 6
Time Frame: at baseline, upon training completion (Week 4), and three months post baseline.
Population: Forty-three caregivers began the study; 42 completed the survey at Month 1; 40 completed the month 3 survey.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 43
Score on a scale
  Baseline | 20.13 (13.27)
  Month 1: number analyzed (Participants) | 42
  Month 1 | 19.70 (12.21)
  Month 3: number analyzed (Participants) | 40
  Month 3 | 16.35 (12.05)

ADVERSE EVENTS:
Time Frame: Data were collected for 3 months.
Arm/Group | Caregivers
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT05996718/Prot_SAP_ICF_000.pdf